CLINICAL TRIAL: NCT01591174
Title: Evaluation of Liquid Gastric Emptying and Plasma Ghrelin in Children With Functional Dyspepsia
Brief Title: Ghrelin and Gastric Emptying in Children With Functional Dyspepsia
Acronym: GHR
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Nadia Hijaz, MD, Fellow, Children's Mercy Hospital, Section of Gastroenterology, Children's Mercy Hospital Kansas City
Other Study IDs: Ghrelin 12010078
Record Dates: First submitted 2012-05-02; First posted 2012-05-03 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia; Postprandial Distress Syndrome; ghrelin; C-13 acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — breath specimen blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Functional Dyspepsia with PDS: Study participants 8-17 years of age will be recruited for this arm after an evaluation at Children's Mercy Hospital and Clinics in the Abdominal Pain Clinic (APC)or in the Section of Gastroenterology, general, and diagnosed with FD, fail to respond to acid suppression therapy and have Postprandial Distress Syndrome (PDS).
- Functional Dyspepsia without PDS: Study participants 8-17 years of age will be recruited for this arm after an evaluation at Children's Mercy Hospital and clinics (CMH) Abdominal Pain Clinic (APC)or the Section of Gastroenterology, general, and diagnosed with FD, fail to respond to acid suppression therapy and do not have Postprandial Distress Syndrome (PDS).
- Control Group: Healthy participants 8-17 years of age recruited from internal advertising within Children's Mercy Hospital and Clinics.

SUMMARY:
The purpose of this research is to see if there are differences between children who have FD and children without FD in the ability of the stomach to empty food and/or in ghrelin hormone levels before and after eating.

Chronic abdominal pain is the most common persistent pain condition in children and adolescents. One of the most often diagnosed types of abdominal pain is functional dyspepsia (FD). FD is abdominal pain or discomfort (e.g., nausea, bloating) in the upper abdomen that does not get better by having a bowel movement.

One possible explanation for having FD is a delay in the emptying of food from the stomach, or delayed gastric (stomach) emptying. Failing to empty the stomach quickly enough may result in the feeling of being full and cause symptoms of bloating, nausea, vomiting and pain. Further, hormonal changes occur before, during, or after eating food that appear to impact stomach emptying.

One of the hormones that changes with meals is called ghrelin. The relationship between ghrelin and stomach emptying needs to be explored more in children with FD. Better understanding of what causes FD symptoms may help us to improve treatment for this condition.

DETAILED DESCRIPTION:
Functional Dyspepsia (FD) is defined as the presence of persistent or recurrent pain or discomfort centered in the upper abdomen with no evidence of organic disease likely to explain the symptoms.

This pain or discomfort must not be exclusively relieved by defecation or associated with the onset of a change in stool frequency or stool form.

Initially, the FD classification criteria included 3 subtypes: ulcer-like, in which pain is the predominant symptom; dysmotility-like, in which discomfort is the predominant symptom; and, unspecified. In 2006, however, the criteria were revised by the Rome III committees. In adults, the previous FD subtypes were eliminated and replaced by two new subtypes: (i) postprandial distress syndrome (PDS), characterized by postprandial fullness or early satiety; and, (ii) epigastric pain syndrome (EPS), characterized by epigastric pain or burning unrelated to meals. In children, the Rome II subtypes were eliminated completely. Although the Rome III subtypes have only been applied within adult criteria, there also appear to be meaningful associations in children with FD which may support their adoption in later revisions of the criteria. Specifically, both inflammation (reflected by mast cell density) and self reported anxiety and depression appear to be uniquely associated with PDS in children.

FD is a common disorder of the upper gastrointestinal (GI) tract, occurring in 26% to 34% of the general population. FD is present in as many as 80% of children being evaluated for chronic abdominal pain. FD is best explained by a biopsychological model with dysfunction within the brain-gut axis. The model suggests that FD is as a result of interaction between biological (e.g., inflammation, mechanical, or sensory dysfunction), psychological (e.g., anxiety, depression, somatization), and social (e.g., interactions with parents, teachers, or peers) factors, which may be interactive with each other. Delayed gastric emptying is one of the mechanical factors which have been implicated. Other mechanisms are visceral hypersensitivity and impaired gastric fundic accommodation.

Delayed gastric emptying has been shown in up to 66% of children with FD. Most of previous studies in children used solid GE as a measure to explain the function of pyloric emptying. However, liquids GE is a good measure to predict the function of fundic accommodation, visceral hypersensitivity as well as pyloric emptying, in which, all these mechanisms were suggested in the mechanical pathophysiological model of FD specifically PDS subtypes. In order to measure gastric emptying (GE), the 13C-acetate breath test (ABT) has the potential to replace 99mtechnetium colloid-based scintigraphy which is the "gold standard" for measuring GE. ABT has an advantage over scintigraphy in that it is a rapid, technically simple, safe and inexpensive means to assess liquid GE in children. As such, it may be more easily utilized as a diagnostic technique in standard clinical practice.

Gastric motility is mainly regulated by extrinsic autonomic nerves, intrinsic neurons of the stomach, and GI hormones. It is hypothesized that these hormones strongly affect hunger and energy expenditure and may be are altered in dyspeptic disorders affecting gastric motility. Because altered gut-brain interactions may underlie symptom generation in FD and ghrelin is an important gut peptide related to the gut-brain axis, plasma concentrations of ghrelin in patients with FD have been investigated in several studies.

Ghrelin is a motilin-related peptide mainly synthesized and released by A-like cells in the stomach. Ghrelin acts as an endogenous ligand of growth hormone secretagogue receptor (GHSR). Ghrelin receptors are present in the anterior pituitary hypothalamus. There are two forms of ghrelin. The first form is acyl ghrelin, comprising 28 amino acid residues with an n-octanoyl ester at Ser3 that is essential for its biologic activity, which acts as an endogenous ligand of growth hormone secretagogue receptor type 1a (GHS-R1a). Acyl ghrelin is easily and rapidly degraded to the second form, desacyl ghrelin, or smaller fragments.

Functionally, ghrelin level progressively rises during fasting to peak just prior to a meal and fall to its lowest level about an hour after eating. Ghrelin level again starts increasing approximately 2 hours after eating to peak again before the next meal. A close relationship has been documented between ghrelin and gastric motility in rats. In humans, it has been demonstrated that ghrelin increases the gastric emptying rate in healthy, but not in obese, controls. Ghrelin has a well-established role in increasing appetite and food intake. These pieces of evidence have led to speculation that altered ghrelin function may contribute to the disturbed gastric motility and appetite loss seen in FD. Moreover, ghrelin agonist administration is found to have stimulatory effect on appetite in FD patients and idiopathic gastroparesis.

Considering that most symptoms of FD are typically related to food intake, postprandial ghrelin level has been investigated in several studies. It has been shown that fasting ghrelin level, in general, is inversely related to gastric emptying time (i,e., lower fasting ghrelin is associated with greater delay in GE). However, this relation is disrupted in FD patients, as these patients do not demonstrate an increase in fasting ghrelin level. Although results have been somewhat conflicting, some previous studies support a role for ghrelin in FD in adults. Takamori et al. reported that fasting desacyl and total ghrelin levels were significantly lower in FD patients than in controls. Further, fasting and postprandial levels were not significantly different in FD, as compared to a significant drop from fasting to postprandial level seen in controls, which suggests that fasting ghrelin does not increase as expected during fasting in FD patients. Consistent with this, Lee et al. showed that delayed GE has been reported in the majority of adults with FD where abnormally low total pre-prandial ghrelin levels were observed. However, the relationship between FD and ghrelin may differ by FD subtype. Shindo et al. reported that fasting acyl ghrelin levels were significantly lower in PDS adult patients than in healthy volunteers. Further, they demonstrated that Tmax value reflective of GE in PDS patients was significantly higher than in healthy volunteers, as measured using the 13-C (carbon) acetate breath test. These results suggested that acyl ghrelin is more biologically important and might play a role in the pathophysiology of the PDS subtype of FD through its effect on gastric emptying.

Collectively, previous studies suggest a relationship between plasma ghrelin concentration and FD, or FD subtype, in adults. Further, it seems likely that this occurs through the impact of ghrelin on gastric emptying in adults. However, to the best of our knowledge, the role of ghrelin in pediatric FD and it its relation to gastric motility in children has not been previously studied. There is a need to investigate the possible role of ghrelin in its two different forms, as well as its relation to gastric motility, in children with FD as a group and across possible subtypes in order to establish better understanding of the pathophysiology of FD. This study may help to build a mechanical pathway model for FD etiology, explore the pharmacokinetics of the ghrelin hormone, and establish its correlation to liquid gastric emptying. If a relationship is established, future work can explore a potential therapeutic role for ghrelin agonist in FD or specific FD subtypes.

ELIGIBILITY:
Inclusion Criteria:

* All: Participants 8-17 years of age
* FD arms: Patients identified in CMH/Abdominal Pain Team Clinic with Functional Dyspepsia who meet exclusion criteria.
* Control arm: healthy participants who meet exclusion criteria.

Exclusion Criteria:

* History of upper gastrointestinal surgery or intestinal obstruction.
* History of disease or symptoms suggestive of underlying malabsorption, Inflammatory Bowel Disease (IBD), or Peptic Ulcer Disease (PUD).
* History or evidence of chronic illness requiring regular medical care such as diabetes mellitis (DM), liver, heart, kidney, endocrine, or pulmonary disease and asthma that precludes accurate exhalation into the study breath collection apparatus.
* Any patient with body Mass index (BMI) less than or equal to 10th percentile for age; or equal to or greater than 90th percentile for age.
* Patient and/or parent not able to read English.
* Current pregnancy.
* History of milk allergy.
* Prokinetic or psychotropic medications used within the last 72 hour prior to study.
* Inability to exhale into study breath collection apparatus as directed.
* Recent acute illness that occurs prior to study visit.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All FD patients will be recruited from the Section of Gastroenterology at the Children's Mercy Hospital and Clinics. The control group will be recruited by advertisement within Children's Mercy Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2016-04-22 (Actual)

PRIMARY OUTCOMES:
Children with FD: exploration of relationships between ghrelin concentration, liquid gastric emptying, and dyspepsia subtype | Duration of 4-hour study visit
  Blood samples will be compared pre/post test meal for FD cohorts (EPS/PDS), controls: 0 time/baseline; 6 times/post meal. Associations between relationship of plasma ghrelin type's (acyl and desacyl) pre and postprandial levels & gastric emptying studied.C-13 acetate to be given and amount of 13CO2 determined for each time point (1 pre/ 14 post meal) using equation nested in software package with UBit IR-300 spectrometer. The concentration of 13CO2 and 12CO2 in the exhaled breath samples to be measured by infrared spectrometry.

SECONDARY OUTCOMES:
Children with FD: SUBJECTIVE SYMPTOM SEVERITY and correlations between plasma ghrelin concentrations (acyl and desacyl) and gastric emptying. | Duration of 4-hour study visit
  Intensity of 5 symptoms associated with FD (burning, nausea, bloating, belching, epigastric pain) will be graded x6 (1 pre and 5 post-meal).

CONTACTS AND LOCATIONS:
Overall Officials: Nadia M Hijaz, MD, Principal Investigator — Fellow, Children's Mercy Hospital, Section of Gastroenterology
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Background] Drossman DA. The functional gastrointestinal disorders and the Rome III process. Gastroenterology. 2006 Apr;130(5):1377-90. doi: 10.1053/j.gastro.2006.03.008. No abstract available. PMID 16678553
- [Background] Suzuki H, Nishizawa T, Hibi T. Therapeutic strategies for functional dyspepsia and the introduction of the Rome III classification. J Gastroenterol. 2006 Jun;41(6):513-23. doi: 10.1007/s00535-006-1847-5. PMID 16868798
- [Background] Akamizu T, Iwakura H, Ariyasu H, Kangawa K. Ghrelin and functional dyspepsia. Int J Pept. 2010;2010:548457. doi: 10.1155/2010/548457. Epub 2010 Jan 12. PMID 20721353
- [Background] Schurman JV, Singh M, Singh V, Neilan N, Friesen CA. Symptoms and subtypes in pediatric functional dyspepsia: relation to mucosal inflammation and psychological functioning. J Pediatr Gastroenterol Nutr. 2010 Sep;51(3):298-303. doi: 10.1097/MPG.0b013e3181d1363c. PMID 20479684
- [Background] Castillo EJ, Camilleri M, Locke GR, Burton DD, Stephens DA, Geno DM, Zinsmeister AR. A community-based, controlled study of the epidemiology and pathophysiology of dyspepsia. Clin Gastroenterol Hepatol. 2004 Nov;2(11):985-96. doi: 10.1016/s1542-3565(04)00454-9. PMID 15551251
- [Background] Drossman DA, Li Z, Andruzzi E, Temple RD, Talley NJ, Thompson WG, Whitehead WE, Janssens J, Funch-Jensen P, Corazziari E, et al. U.S. householder survey of functional gastrointestinal disorders. Prevalence, sociodemography, and health impact. Dig Dis Sci. 1993 Sep;38(9):1569-80. doi: 10.1007/BF01303162. PMID 8359066
- [Background] Schurman JV, Friesen CA, Danda CE, Andre L, Welchert E, Lavenbarg T, Cocjin JT, Hyman PE. Diagnosing functional abdominal pain with the Rome II criteria: parent, child, and clinician agreement. J Pediatr Gastroenterol Nutr. 2005 Sep;41(3):291-5. doi: 10.1097/01.mpg.0000178438.64675.c4. PMID 16131983
- [Background] Hyams JS, Hyman PE. Recurrent abdominal pain and the biopsychosocial model of medical practice. J Pediatr. 1998 Oct;133(4):473-8. doi: 10.1016/s0022-3476(98)70053-8. No abstract available. PMID 9787683
- [Background] Takamori K, Mizuta Y, Takeshima F, Akazawa Y, Isomoto H, Ohnita K, Ohba K, Omagari K, Shikuwa S, Kohno S. Relation among plasma ghrelin level, gastric emptying, and psychologic condition in patients with functional dyspepsia. J Clin Gastroenterol. 2007 May-Jun;41(5):477-83. doi: 10.1097/01.mcg.0000225614.94470.47. PMID 17450030
- [Background] Ogiso K, Asakawa A, Amitani H, Inui A. Ghrelin: a gut hormonal basis of motility regulation and functional dyspepsia. J Gastroenterol Hepatol. 2011 Apr;26 Suppl 3:67-72. doi: 10.1111/j.1440-1746.2011.06630.x. PMID 21443713
- [Background] Riezzo G, Chiloiro M, Guerra V, Borrelli O, Salvia G, Cucchiara S. Comparison of gastric electrical activity and gastric emptying in healthy and dyspeptic children. Dig Dis Sci. 2000 Mar;45(3):517-24. doi: 10.1023/a:1005493123557. PMID 10749327
- [Background] Heyman S. Gastric emptying in children. J Nucl Med. 1998 May;39(5):865-9. PMID 9591590
- [Background] Hou XH, Li Q, Zhu L, Xie X, Chen JD. Correlation of gastric liquid emptying with various thresholds of sensation in healthy controls and patients with functional dyspepsia. Dig Dis Sci. 2004 Feb;49(2):188-95. doi: 10.1023/b:ddas.0000017437.20932.8b. PMID 15104356
- [Background] Maes BD, Ghoos YF, Geypens BJ, Hiele MI, Rutgeerts PJ. Relation between gastric emptying rate and energy intake in children compared with adults. Gut. 1995 Feb;36(2):183-8. doi: 10.1136/gut.36.2.183. PMID 7883214
- [Background] Jones BL, Pearce RE, Abdel-Rahman SM, Friesen CA, James LP, Kearns GL. Characterization of delayed liquid gastric emptying in children by the (13)C-acetate breath test. J Breath Res. 2009 Dec;3(4):047004. doi: 10.1088/1752-7155/3/4/047004. Epub 2009 Nov 27. PMID 21386201
- [Background] Braden B, Adams S, Duan LP, Orth KH, Maul FD, Lembcke B, Hor G, Caspary WF. The [13C]acetate breath test accurately reflects gastric emptying of liquids in both liquid and semisolid test meals. Gastroenterology. 1995 Apr;108(4):1048-55. doi: 10.1016/0016-5085(95)90202-3. PMID 7698571
- [Background] Hauser B, De Schepper J, Caveliers V, Salvatore S, Salvatoni A, Vandenplas Y. Variability of the 13C-acetate breath test for gastric emptying of liquids in healthy children. J Pediatr Gastroenterol Nutr. 2006 Apr;42(4):392-7. doi: 10.1097/01.mpg.0000215306.40546.17. PMID 16641577
- [Background] Barbosa L, Vera H, Moran S, Del Prado M, Lopez-Alarcon M. Reproducibility and reliability of the 13C-acetate breath test to measure gastric emptying of liquid meal in infants. Nutrition. 2005 Mar;21(3):289-94. doi: 10.1016/j.nut.2004.05.027. PMID 15797668
- [Background] Gatti C, di Abriola FF, Dall'Oglio L, Villa M, Franchini F, Amarri S. Is the 13C-acetate breath test a valid procedure to analyse gastric emptying in children? J Pediatr Surg. 2000 Jan;35(1):62-5. doi: 10.1016/s0022-3468(00)80015-9. PMID 10646776
- [Background] Ueno H, Shiiya T, Nakazato M. Translational research of ghrelin. Ann N Y Acad Sci. 2010 Jul;1200:120-7. doi: 10.1111/j.1749-6632.2010.05509.x. PMID 20633140
- [Background] Chanoine JP. Ghrelin in growth and development. Horm Res. 2005;63(3):129-38. doi: 10.1159/000084688. Epub 2005 Mar 24. PMID 15795510
- [Background] Tack J, Depoortere I, Bisschops R, Delporte C, Coulie B, Meulemans A, Janssens J, Peeters T. Influence of ghrelin on interdigestive gastrointestinal motility in humans. Gut. 2006 Mar;55(3):327-33. doi: 10.1136/gut.2004.060426. Epub 2005 Oct 10. PMID 16216827
- [Background] Lee KJ, Cha DY, Cheon SJ, Yeo M, Cho SW. Plasma ghrelin levels and their relationship with gastric emptying in patients with dysmotility-like functional dyspepsia. Digestion. 2009;80(1):58-63. doi: 10.1159/000215389. Epub 2009 Jun 3. PMID 19494492
- [Background] Shindo T, Futagami S, Hiratsuka T, Horie A, Hamamoto T, Ueki N, Kusunoki M, Miyake K, Gudis K, Tsukui T, Iwakiri K, Sakamoto C. Comparison of gastric emptying and plasma ghrelin levels in patients with functional dyspepsia and non-erosive reflux disease. Digestion. 2009;79(2):65-72. doi: 10.1159/000205740. Epub 2009 Feb 27. PMID 19246923
- [Background] Fukuda H, Mizuta Y, Isomoto H, Takeshima F, Ohnita K, Ohba K, Omagari K, Taniyama K, Kohno S. Ghrelin enhances gastric motility through direct stimulation of intrinsic neural pathways and capsaicin-sensitive afferent neurones in rats. Scand J Gastroenterol. 2004 Dec;39(12):1209-14. PMID 15742997
- [Background] Trudel L, Tomasetto C, Rio MC, Bouin M, Plourde V, Eberling P, Poitras P. Ghrelin/motilin-related peptide is a potent prokinetic to reverse gastric postoperative ileus in rat. Am J Physiol Gastrointest Liver Physiol. 2002 Jun;282(6):G948-52. doi: 10.1152/ajpgi.00339.2001. PMID 12016119
- [Background] Heath RB, Jones R, Frayn KN, Robertson MD. Vagal stimulation exaggerates the inhibitory ghrelin response to oral fat in humans. J Endocrinol. 2004 Feb;180(2):273-81. doi: 10.1677/joe.0.1800273. PMID 14765979
- [Background] Lin Z, Eaker EY, Sarosiek I, McCallum RW. Gastric myoelectrical activity and gastric emptying in patients with functional dyspepsia. Am J Gastroenterol. 1999 Sep;94(9):2384-9. doi: 10.1111/j.1572-0241.1999.01362.x. PMID 10483996
- [Background] Valera Mora ME, Scarfone A, Valenza V, Calvani M, Greco AV, Gasbarrini G, Mingrone G. Ghrelin does not influence gastric emptying in obese subjects. Obes Res. 2005 Apr;13(4):739-44. doi: 10.1038/oby.2005.83. PMID 15897483
- [Background] Wren AM, Bloom SR. Gut hormones and appetite control. Gastroenterology. 2007 May;132(6):2116-30. doi: 10.1053/j.gastro.2007.03.048. PMID 17498507
- [Background] Akamizu T, Iwakura H, Ariyasu H, Hosoda H, Murayama T, Yokode M, Teramukai S, Seno H, Chiba T, Noma S, Nakai Y, Fukunaga M, Nakai Y, Kangawa K; FD Clinical Study Team. Repeated administration of ghrelin to patients with functional dyspepsia: its effects on food intake and appetite. Eur J Endocrinol. 2008 Apr;158(4):491-8. doi: 10.1530/EJE-07-0768. PMID 18362296
- [Background] Ejskjaer N, Dimcevski G, Wo J, Hellstrom PM, Gormsen LC, Sarosiek I, Softeland E, Nowak T, Pezzullo JC, Shaughnessy L, Kosutic G, McCallum R. Safety and efficacy of ghrelin agonist TZP-101 in relieving symptoms in patients with diabetic gastroparesis: a randomized, placebo-controlled study. Neurogastroenterol Motil. 2010 Oct;22(10):1069-e281. doi: 10.1111/j.1365-2982.2010.01519.x. Epub 2010 Jun 28. PMID 20524987
- [Background] Tack J, Depoortere I, Bisschops R, Verbeke K, Janssens J, Peeters T. Influence of ghrelin on gastric emptying and meal-related symptoms in idiopathic gastroparesis. Aliment Pharmacol Ther. 2005 Nov 1;22(9):847-53. doi: 10.1111/j.1365-2036.2005.02658.x. PMID 16225494
- [Background] Ang D, Nicolai H, Vos R, Mimidis K, Akyuz F, Kindt S, Vanden Berghe P, Sifrim D, Depoortere I, Peeters T, Tack J. Influence of ghrelin on the gastric accommodation reflex and on meal-induced satiety in man. Neurogastroenterol Motil. 2009 May;21(5):528-33, e8-9. doi: 10.1111/j.1365-2982.2008.01239.x. Epub 2008 Jan 30. PMID 19210631
- [Background] Nishizawa T, Suzuki H, Nomoto Y et al. Enhanced plasma ghrelin levels in patients with functional dyspepsia. Aliment. Pharmacol. Ther. 2006; 24 (Suppl. 4): 104-10. 02.01.12